CLINICAL TRIAL: NCT00411931
Title: A Clinical Investigation of the Pharmacokinetics and Safety of MultiHance in Patients From 2-5 Years of Age Undergoing A Clinical Indicated MRI of the CNS
Brief Title: A Pharmacokinetics Study of MultiHance in Pediatric Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Gianpaolo Pirovano, MD, Executive Director, Corporate Medical Development, Bracco Diagnostics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MH 119
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Central Nervous System Pathology
MeSH Terms: interventions — gadobenic acid

INTERVENTIONS:
Drug: Multihance — 0.5M administered as a single injection

SUMMARY:
Compare relative exposure in the younger age group in order to supplement the PK profile already determined in older children and adults

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 2 and 5 years of age
* Obtained informed consent from patient's parent or guardian
* Obtain assent when applicable according to local law
* Known or suspected disease of the central nervous system (brain or spine)
* Referred for MRI of the brain or spine requiring an injection of an MR contrast agent

Exclusion Criteria:

* Contraindications to MR examination
* Undergoing MRI in an emergency situation
* Known allergy to one or more ingredients in the contrast agent or history of hypersensitivity to gadolinium or metals
* Sickle cell anemia
* Likely to undergo an invasive examination within 72 hours after administration of the investigational product

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Assess the blood PK of Multihance in patients from 2 to 5 years of age | up to 24 hours post dose

SECONDARY OUTCOMES:
Evaluate the safety of Multihance in patients from 2 to 5 years of age | through 72 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, M. D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Krakow, Poland